CLINICAL TRIAL: NCT02186678
Title: Comparison of Diagnostic Performances of 68Ga-DOTATATE PET-CT and 18F-FDOPA PET-CT in Paragangliomas and Pheochromocytomas Evaluation: Monocentric Prospective Study
Brief Title: Comparison of Diagnostic Performances of 68Ga-DOTATATE PET-CT and 18F-FDOPA PET-CT in Paragangliomas and Pheochromocytomas Evaluation
Acronym: DOTATATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-26
Record Dates: First submitted 2014-06-04; First posted 2014-07-10 (Estimated); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Paragangliomas; Pheochromocytomas
MeSH Terms: conditions — Paraganglioma; Pheochromocytoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- assesment by 68Ga-DOTATATE PET-CT (Experimental)
  Interventions: Other: PET-CT

INTERVENTIONS:
Other: PET-CT

SUMMARY:
18F-FDOPA PET-CT is currently the gold standard in the evaluation of Pheochromocytomas and Paragangliomas (PHEO - PGL) since these tumors can also decarboxylate amino acids such as dihydroxyphenylalanine (DOPA). This property is common to tumors of the APUD system (Amine Precursor Uptake and Decarboxylation). In recent years, PET (Positron Emission Tomography) imaging using peptide receptors has gained an increasing role in the management of NETs. The use of somatostatin agonists, radiolabeled with gallium-68 (68Ga) enables targeting of Somatostatin receptors (SSTRs) with a PET resolution. This has improved diagnosis of SSTRs-expressing tumors, including PGLs.

In the present study, the investigators have chosen DOTATATE (Nal3-octreotate) rather than other agonists (DOTATOC and DOTANOC), because of its higher affinity for SST2 which is the most overexpressed subtype in PHEO/PGL. However, performances of 18F-FDOPA PET-CT and 68Ga-DOTATATE PET-CT have never been compared in this clinical setting.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18

* PHEO or PGL: initial staging or restaging
* Reference imaging within the last 2 months: multiphasic cervico-thoracoabdominal CT scan, 18F-FDOPA PET-CT and head and neck MRI (if head and neck localization

Exclusion Criteria:

Pregnant or breast-feeding woman

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-07-18 (Actual); Primary Completion 2015-10-05 (Actual); Study Completion 2023-04-05 (Actual)

PRIMARY OUTCOMES:
interest of the the contribution of 68Ga-DOTATATE PET-CT in the staging of PHEO/PGL | 7 months
  The primary outcome measure is to determine the contribution of 68Ga-DOTATATE PET-CT in the staging of PHEO/PGL. We will document the number of additional foci detected by 68Ga-DOTATATE PET-CT compared to 18F-FDOPA PET-CT.

SECONDARY OUTCOMES:
assesment of 68Ga-DOTATATE PET-CT to anatomical imaging | 7 months
  The secondary objective is to compare , to assess the factors influencing its sensitivity concerning the tumor location

OTHER OUTCOMES:
assesment of 68Ga-DOTATATE PET-CT to anatomical imaging | 7 months
  The third objective is to compare 68Ga-DOTATATE PET-CT to anatomical imaging, to assess the factors influencing its sensitivity concerning the genetic status,
assesment of 68Ga-DOTATATE PET-CT to anatomical imaging | 7 months
  The fourth objective is to compare 68Ga-DOTATATE PET-CT to anatomical imaging, to assess the factors influencing its sensitivity concerning Somatostatin receptor expression

CONTACTS AND LOCATIONS:
Overall Officials: David TAIEB, MD, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France